CLINICAL TRIAL: NCT02347462
Title: A Prospective Open Randomized Clinical Trial Comparing Bilevel Positive Airway Pressure (BiPAP) Therapy Against Standard Therapy for Children Hospitalized With an Acute Exacerbation of Asthma Unresponsive to Inhaled Bronchodilators.
Brief Title: Bilevel Positive Airway Pressure (BiPAP) for the Treatment of Moderate to Severe Acute Asthma Exacerbations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: we were not able to work through the logistics of the study to support enrolment in ER
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Seear, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H14-02397
Record Dates: First submitted 2015-01-14; First posted 2015-01-27 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Asthma; Status Asthmaticus
Keywords: BiPAP
MeSH Terms: conditions — Asthma; Status Asthmaticus | interventions — Continuous Positive Airway Pressure; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BiPAP plus standard care (Experimental): Bilevel Positive Airway Pressure (BiPAP) plus standard care according to the hospital's severe asthma protocol
  Interventions: Device: Bilevel Positive Airway Pressure (BiPAP) (Trilogy BiPAP, Philips Respironics); Other: Standard care
- Standard care alone (Active Comparator): Standard care according to the hospital's severe asthma protocol
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Bilevel Positive Airway Pressure (BiPAP) (Trilogy BiPAP, Philips Respironics) — Children in the intervention group will receive BiPAP (Trilogy, Philips Respironics; spontaneous trigger mode) via a nasal or full face mask. End expiratory positive airway pressure (EPAP) will be set at 5cm H20. Inspiratory positive airway pressure (IPAP) will be titrated to achieve a tidal volume of 6 - 9 ml/kg. These settings will remain unchanged throughout the study period.
  Other Names: Trilogy BiPAP, Philips Respironics
  Arms: BiPAP plus standard care
Other: Standard care — Standard care according to the hospital severe asthma protocol

SUMMARY:
Bilevel Positive Airway Pressure (BiPAP) is increasingly being reported as an effective and safe method of respiratory support for children with severe asthma exacerbations unresponsive to standard therapies and with impending respiratory failure. Much of the evidence base supporting its use comes from retrospective observational studies, and there is currently a lack of data from randomized controlled trials to inform this practice.

The investigators hypothesize that the use of BiPAP in children with moderate to severe asthma exacerbations could reduce the length of hospital stay, need for invasive ventilation, and use of intravenous bronchodilators. The investigators aim to test this hypothesis by randomizing children attending the Emergency Department with a moderate to severe clinical severity score refractory to inhaled bronchodilators to receive either BiPAP in addition to standard asthma care, or standard care alone.

DETAILED DESCRIPTION:
Children aged 2 - 18 years presenting to the Emergency Department (ED) with a moderate or severe asthma exacerbation (Pediatric Respiratory Assessment Measure (PRAM) of > 3) who fail to improve clinically with standard ED management with inhaled salbutamol and ipratropium will be randomized to receive either standard asthma management according to our local severe asthma guideline or management with BiPAP in addition to standard care. Both groups will receive a comparable dose of systemic steroid and hourly salbutamol inhalers with subsequent weaning according to PRAM score. Patients randomized to receive BiPAP will be admitted to the Pediatric Intensive Care Unit (PICU) and those randomized to the control group will be admitted to the medical ward. Both groups will be monitored with 3-hourly PRAM scoring through the duration of their admission.

ELIGIBILITY:
Inclusion Criteria:

* 2-18 years old
* Admitted to BC Children's Hospital with a clinical diagnosis of an acute asthma exacerbation
* PRAM score of >3 following initial treatment with three rounds of inhaled salbutamol and ipratropium bromide, and one dose of systemic steroid
* Parents willing and able to sign consent
* Children over the age of 6 willing to provide assent

Exclusion Criteria:

* Clinical suspicion of co-existing bacterial pneumonia: focal crackles or bronchial breathing, and/or major chest x-ray findings
* Impending respiratory failure at presentation requiring direct PICU admission
* Receiving maintenance dose of oral steroid at time of hospital admission
* Any contraindication to BiPAP use including altered mental status, recent bowel surgery, intractable vomiting, or inability to protect airway
* Current tracheostomy, home ventilation (IPPV or NIPPV) or home oxygen requirement
* History of congenital heart disease or chronic respiratory disease (including bronchopulmonary dysplasia, cystic fibrosis, pulmonary hypertension)
* Craniofacial abnormality precluding the use of a tight fitting facial mask

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pediatric Respiratory Assessment Measure (PRAM) clinical severity score of ≤ 3 (mild) | Assessed at initiation, and 3-hourly thereafter until hospital discharge (an estimated average duration of 4 days)
  PRAM score includes assessment of oxygen saturations, suprasternal retractions, scalene muscle contraction, air entry and wheezing.

SECONDARY OUTCOMES:
Intubation and complication rates | Patients will be followed for the duration of their hospital stay (an estimated average of 4 days) with data collection relative to this outcome on a daily basis
  Number of children in each arm requiring intubation and mechanical ventilation, and experiencing significant treatment-related side effects
Hospital re-admission | Within 48 hours of initial hospital discharge
  Number of children in each arm failing initial hospital discharge and requiring re-admission within 48 hours
Inhaled bronchodilator utilization | Patients will be followed for the duration of their hospital stay (an estimated average of 4 days) with data collection relative to this outcome on a daily basis
  Comparison of the median daily dose of inhaled salbutamol received by children in each arm,
Intravenous bronchodilator utilization | Patients will be followed for the duration of their hospital stay (an estimated average of 4 days) with data collection relative to this outcome on a daily basis
  Comparison of the total number of hours of intravenous bronchodilator infusions received by children in each arm
Length of hospital stay | Length of stay will be calculated at the time of each child's hospital discharge (estimated 4 days after hospital admission and recruitment to study)
  Duration of time from hospital admission to the patient meeting hospital discharge criteria

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seear, MD, Principal Investigator — University of British Columbia
Locations (1):
- Children's and Women's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Martinez FD, Vercelli D. Asthma. Lancet. 2013 Oct 19;382(9901):1360-72. doi: 10.1016/S0140-6736(13)61536-6. Epub 2013 Sep 13. PMID 24041942
- [Background] Papiris SA, Manali ED, Kolilekas L, Triantafillidou C, Tsangaris I. Acute severe asthma: new approaches to assessment and treatment. Drugs. 2009;69(17):2363-91. doi: 10.2165/11319930-000000000-00000. PMID 19911854
- [Background] Soroksky A, Klinowski E, Ilgyev E, Mizrachi A, Miller A, Ben Yehuda TM, Shpirer I, Leonov Y. Noninvasive positive pressure ventilation in acute asthmatic attack. Eur Respir Rev. 2010 Mar;19(115):39-45. doi: 10.1183/09059180.00006109. PMID 20956164
- [Background] Meduri GU, Cook TR, Turner RE, Cohen M, Leeper KV. Noninvasive positive pressure ventilation in status asthmaticus. Chest. 1996 Sep;110(3):767-74. doi: 10.1378/chest.110.3.767. PMID 8797425
- [Background] Thill PJ, McGuire JK, Baden HP, Green TP, Checchia PA. Noninvasive positive-pressure ventilation in children with lower airway obstruction. Pediatr Crit Care Med. 2004 Jul;5(4):337-42. doi: 10.1097/01.pcc.0000128670.36435.83. PMID 15215002
- [Background] Basnet S, Mander G, Andoh J, Klaska H, Verhulst S, Koirala J. Safety, efficacy, and tolerability of early initiation of noninvasive positive pressure ventilation in pediatric patients admitted with status asthmaticus: a pilot study. Pediatr Crit Care Med. 2012 Jul;13(4):393-8. doi: 10.1097/PCC.0b013e318238b07a. PMID 22067982
- [Background] Ducharme FM, Chalut D, Plotnick L, Savdie C, Kudirka D, Zhang X, Meng L, McGillivray D. The Pediatric Respiratory Assessment Measure: a valid clinical score for assessing acute asthma severity from toddlers to teenagers. J Pediatr. 2008 Apr;152(4):476-80, 480.e1. doi: 10.1016/j.jpeds.2007.08.034. Epub 2007 Oct 31. PMID 18346499